CLINICAL TRIAL: NCT00038961
Title: A Multicenter, Randomized, Double-blind, Parallel Group Trial to Demonstrate the Efficacy of Fondaparinux Sodium in Association With Intermittent Pneumatic Compression (IPC) Versus IPC Used Alone for the Prevention of Venous Thromboembolic Events in Subjects at Increased Risk Undergoing Major Abdomi
Brief Title: A Study to Evaluate the Efficacy and Safety of Fondaparinux Sodium When Used With Intermittent Pneumatic Compression to Prevent Venous Thromboembolic (IPC) Versus IPC Alone for the Prevention of Venous Thromboembolic Events in Subjects at Increased Risk Undergoing Major Abdominal Surgery (APOLLO).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 103414
Record Dates: First submitted 2002-06-05; First posted 2002-06-10 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Thromboembolism
Keywords: fondaparinux sodium; DVT Prevention; abdominal surgery; VTE prevention; venous thromboembolism; pulmonary embolism
MeSH Terms: conditions — Thromboembolism; Venous Thromboembolism; Pulmonary Embolism | interventions — Fondaparinux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + intermittent pneumatic compression (IPC) (Placebo Comparator)
  Interventions: Other: placebo
- fondaparinux + intermittent pneumatic compression (IPC) (Experimental)
  Interventions: Drug: fondaparinux sodium

INTERVENTIONS:
Drug: fondaparinux sodium — 2.5 mg fondparinux sodium, daily, s.c. starting 6 to 8 hours after surgical closure for up to 7 +/- 2 days, administered on top of IPC +/- elastic stockings (ES)
  Arms: fondaparinux + intermittent pneumatic compression (IPC)
Other: placebo — placebo, daily, s.c. starting 6 to 8 hours after surgical closure for up to 7 +/- 2 days, administered on top of IPC +/- elastic stockings (ES)
  Arms: Placebo + intermittent pneumatic compression (IPC)

SUMMARY:
This is a multicentre, randomized, double-blind, placebo controlled study. During this study all the patients will receive background venous thromboembolism (VTE) mechanical prophylaxis with intermittent pneumatic compression (IPC).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of fondaparinux in the prevention of venous thromboembolism (VTE) in subjects undergoing abdominal surgery at increased risk for VTE. During this study all subjects were to receive background VTE prophylaxis with intermittent pnuematic compression (IPC) ± elastic stockings (ES).

Screening Period ( Day -30-Day 0) all subjects at increased risk of VTE undergoing abdominal surgery and fulfilled the study entry criteria were eligible for the study.

Treatment Period (Day 7 ±2): At the baseline assessment on the day of surgery (Day 1) subjects who satisfied all inclusion/exclusion criteria were randomized (1:1) to receive either fondaparinux or placebo. All the subjects were to receive background therapy with IPC ±ES. The first administration of either fondaparinux 2.5mg or placebo was to take place 6 to 8 hours after surgical closure provided hemostasis was achieved. Thereafter a once daily subcutaneous injection of either fondaparinux 2.5mg or placebo was to be administered up to Day 7 ±2. During the treatment phase, subjects were assessed daily. A mandatory venogram was performed between Day 5 and 10 or earlier in the case of symptomatic VTE, but not more than 1 calendar day after the last study treatment administration.

Follow up Period (Day 30 ±2): A follow-up visit or contact was to take place at Day 30 ±2 days. Use of antithrombotic therapy for prevention of VTE after the mandatory venographyand during the entire Follow-up Period was left to the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing abdominal surgery (any surgery between the diaphragm and pelvic floor) lasting longer than 45 minutes (duration from anesthesia induction to surgical closure)
* Over 40 years of age
* Subject who had signed the informed consent.

Exclusion Criteria:

* Active, clinically significant bleeding
* Documented congenital or acquired bleeding tendency/disorders
* Active ulcerative gastrointestinal disease unless the reason for the present surgery.
* Recent intracranial hemorrhage or recent (less than 3 months prior to randomisation) brain, spinal, or ophthalmologic surgery.
* Indwelling intrathecal or epidural catheters for more than 6 hours after surgical closure.
* Subjects who had a traumatic puncture or unusual difficulty in applying the catheter
* Known cerebral metastasis,
* Subjects in whom hemostasis had not been established 6 hours after surgical closure,
* Current thrombocytopenia,
* Bacterial endocarditis
* Creatinine level above 2.0 mg/dL (180 μmol/L) in a well-hydrated subject,
* Documented hypersensitivity to contrast media,
* Use of any contraindicated drug that could not be combined with the injection of contrast medium,
* Patent with evidence of leg ischemia caused by peripheral vascular disease, unable to undergo IPC and unable to wear Elastic Stockings.

Exclusion criteria related to trial methodology:

* Mental disorders that could interfere with study participation and/or failure to give written informed consent to take part in the study,
* Subject's life expectancy < 6 months,
* Clinical sign of DVT and/or history of recent DVT,
* Participation in any other therapeutic drug study or a device study evaluating DVT prophylaxis within 90 days preceding inclusion,
* Previous participation in a study of fondaparinux sodium,
* Known hypersensitivity to fondaparinux and its excipients,
* Current addictive disorders that could interfere with study participation,
* Administration of heparin, heparinoids, LMWH, oral anticoagulants, dextrans, hirudin, fibrinolytic agents or drugs blocking glycoprotein platelet receptors (GPIIb-IIIa) during the screening period, i.e., from admission to surgery,
* Subjects for whom anticoagulant therapy was contraindicated or who had, due to concomitant disease, an indication for oral anticoagulant or heparins (including LMWH) and who could not discontinue those treatments,
* Women of child-bearing potential: women not using an appropriate contraceptive method during the whole duration of study participation ,
* Subject with body weight <50 kg,
* Subjects, who in the opinion of the investigator, required a pharmacological prophylaxis in addition to intermittent pneumatic compression,
* Known pregnancy and / or women who intended to breastfeed,
* Subjects undergoing vascular surgery such as aorto-femoral bypass graft

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1309 (Actual)
Dates: Start 2001-11; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism (VTE) | adjudicated mandatory venogram positive for DVT between day 5 and day 10; up to day 10 for symptomatic DVT and/or adjudicated non fatal Pe , adjudicated fatal PE
  the incidence of VTE determined as any of the following VTE outcomes recorded up to the first venogram performed or up to Day 10, whichever occurred first: adjudicated manadatory veongram positive for DVT between Day 5 and Day 10; adjudicated symptomatic DVT and/or adjudicated non-fatal PE; adjudicated fatal PE
major bleeding | first study drug injection to 2 days after last study drug injection and first study drug injection up to Day 32
  adjudicated major bleeding

SECONDARY OUTCOMES:
deep vein thrombosis (DVT) | up to Day 10
  Incidence of any DVT, any proximal DVT, and distal only DVT
symptomatic VTE (venous thromboembolism) | up to Day 10 and up to Day 32
  Incidence of adjudicated symptomatic VTE (DVT, non fatal pulmonary embolism (PE), and fatal PE)
initiation of curative treatment | 3 years
  Initiation of curative treatment after VTE assessment used for the primary endpoint evaluation
any VTE and all deaths | up to Day 10
  incidence of any VTE and all deaths
symptomatic VTE and all deaths | up to Day 32
  incidence of adjudicated symptomatic VTE and all deaths
minor bleeding | treatment period and up to day 32
  adjudicated minor bleeding
All major or minor bleeding | 3 years
  All adjudicated (major or minor) bleeding
Adverse events | 3 years
  Adverse Events (AEs/serious adverse events (SAEs))
Transfusion | 3 years
  the need for transfusion and total blood units transfused
Lab parameters | 3 years
  changes from baseline in laboratory parameters
Death | 3 years
  Death

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Turpie AG, Bauer KA, Caprini JA, Comp PC, Gent M, Muntz JE; Apollo Investigators. Fondaparinux combined with intermittent pneumatic compression vs. intermittent pneumatic compression alone for prevention of venous thromboembolism after abdominal surgery: a randomized, double-blind comparison. J Thromb Haemost. 2007 Sep;5(9):1854-61. doi: 10.1111/j.1538-7836.2007.02657.x. PMID 17723125
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103414 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register